CLINICAL TRIAL: NCT02281240
Title: Pathogenesis, Diagnosis, Management and Outcome of Hemostatic Complications in Hematopoietic Stem Cell Transplantation: A Prospective Study
Brief Title: Hemostatic Complications in Hematopoietic Stem Cell Transplantation
Acronym: HCIHSCT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Other Study IDs: Soochowhy 2014
Record Dates: First submitted 2014-10-20; First posted 2014-11-03 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Hemostatic Disorders
Keywords: Hematopoietic Stem Cell Transplantation
MeSH Terms: conditions — Hemostatic Disorders | interventions — Thrombopoietin; Interleukin-11; Heparin

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- With hemostatic complications: The hemostatic and antithrombotic (thrombopoietin, interleukin-11, heparin) measures during HSCT.
  Interventions: Drug: thrombopoietin, interleukin-11, heparin,

INTERVENTIONS:
Drug: thrombopoietin, interleukin-11, heparin, — The hemostatic and antithrombotic (thrombopoietin, interleukin-11, heparin) measures during HSCT.
  Other Names: TPO, IL-11

SUMMARY:
Hemostatic disorders are common and potentially fatal complications in patients undergoing hematopoietic stem-cell transplantation (HSCT). Limited data exist on early diagnosis and prevention of these complications. The investigators undertook this prospective study to determine the incidence, predictor factors, specific pathogenesis, management and survival specially for patients with thrombotic and bleeding complication to better improve outcomes.

DETAILED DESCRIPTION:
Hematopoietic stem cell transplantation（HSCT）is a curative treatment for a variety of malignant and refractory benign hematologic disease, but is associated with life-threatening complications in the same time, among them, hemostatic disorders are not uncommon and presenting an increasing morbidity and mortality in HSCT recipients. Bleeding and thrombosis, two of controversial disorders, have been posing a great threat to patients in the setting of transplantation, and early hemorrhagic complication after HCST is more frequent and subject to more concern by clinical physicians, previous studies have shown the risk of bleeding in HSCT recipients is more than 10-fold higher than neoplastic patients receiving chemotherapy. Meanwhile, thrombosis events, which is characterized by hepatic veno-occlusive diseases (HVOD), transplantation related thrombotic microangiopathy (TA-TMA), and venous thromboembolism (VTE) can not be imprudently ignored with its fatal threat to patients.

Over the last two decades, it has been recognized that the relatively increasing incidence of bleeding and thrombotic complications correlating to the prognosis and quality of life for HSCT recipients. Previous studies have shown that conventional risk factors including graft-versus-host disease (GVHD), infection, thrombocytopenia, the anticoagulation therapy, damage of endothelial cell and conditioning regimen can contribute to the onset of hemostatic disorders in HSCT recipients or can even exacerbate the process. Nevertheless, their roles and detailed pathogenesis in the development of bleeding and thrombosis remain undefined and limited data in Asian population was known about the competing risks of thrombosis and bleeding.

Given the current understanding of hemostatic complication and many unknown mechanisms of relation between thrombosis and hemostasis，we undertook this prospective study to determine the incidence, predictor factors, specific pathogenesis, and survival specially for patients with thrombotic and bleeding complication to better improve outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients signed their informed consents are enrolled; 2. Patients suffering from hematological diseases and undergoing hematopoietic stem cell transplantation.

Exclusion Criteria:

* 1. Patients who have not signed their informed consents; 2. Patients with previous history of platelet disorder or bleeding diathesis; 3. Patients with inadequate renal function or hepatic function, or other essential organ damage.

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The incidence and severity of hemostatic complications in patients following HSCT.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of hemostatic complications in patients following HSCT. | Two years after HSCT

SECONDARY OUTCOMES:
The severity of hemostatic complications in patients following HSCT. | Two years after HSCT
The survival rates of patients with hemostatic complications following HSCT. | Two years after HSCT

CONTACTS AND LOCATIONS:
Overall Officials: Jia Chen, Doctor, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China